CLINICAL TRIAL: NCT07316296
Title: Pharmacologically Modulating the Noradrenergic Arousal System to Reduce Freezing of Gait in Parkinson's Disease: a Multi-centre and Multi-modal Approach
Acronym: AnTi-FREEZE
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: University of Waterloo (Other); Macquarie University, Australia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: R0007688A
Record Dates: First submitted 2025-12-16; First posted 2026-01-05 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Parkinson's Disease (PD); Freezing of Gait; Freezing of Gait Symptoms in Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Atomoxetine Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Atomoxetine in visit 2 and placebo in visit 3 (Experimental)
  Interventions: Drug: Atomoxetine; Drug: Placebo
- Placebo in visit 2 and atomoxetine in visit 3 (Experimental)
  Interventions: Drug: Atomoxetine; Drug: Placebo

INTERVENTIONS:
Drug: Atomoxetine — Single dose, 40mg atomoxetine, capsule
Drug: Placebo — Single dose, placebo (microcrystalline cellulose), capsule

SUMMARY:
The goal of this clinical trial is to learn if the medication atomoxetine can reduce freezing of gait in people with Parkinson's disease. The main questions it aims to answer is:

Does atomoxetine reduce the frequency or severity of freezing of gait? What role does noradrenaline play in freezing of gait?

Researchers will compare atomoxetine to a placebo to see if atomoxetine can improve freezing of gait in people with Parkinson's disease.

Participants will:

Visit the study site for measurements Take atomoxetine or placebo Perform walking assessments and undergo MRI Complete questionnaires about anxiety, stress, and quality of life

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older;
* Diagnosis of idiopathic PD according to MDS Diagnostic Criteria;
* Stabilised on optimal dopaminergic PD treatment for a minimum of four weeks prior to the baseline visit (Visit 1) and for the duration of the trial;
* Presence of FOG symptoms on a daily basis;
* Ability to walk for 10-meters unaided in the dopaminergic ON-state;
* Ability to provide written informed consent in accordance with ICH-GCP and local regulations;
* Willing and able to undergo all clinical trial assessments.

Exclusion Criteria:

* Current and/or previous (within 3 months) participation in a clinical trial;
* Any contra-indications for undergoing MRI-scanning (e.g. claustrophobia or metal parts within the body such as DBS, an infusion pump or a pacemaker);
* Co-morbidity that significantly impacts ambulation (e.g. orthopaedic or rheumatological ailments);
* Severe cognitive impairment hampering the ability to comply with the study protocol;
* Active psychosis that would impact the ability to comply with the study protocol;
* Severe cardiovascular disorders: severe hypertension (Sustained (Sitting) hypertension of ≥180 mmHg systolic or ≥110 mmHg diastolic, defined by the average of three observations, each at least 3 minutes apart, with the participant having assumed the required position for at least 3 minutes), heart failure, arterial occlusive disease, angina, haemodynamically significant congenital heart disease, cardiomyopathies, myocardial infarction, potentially life-threatening arrhythmias, long QT interval syndrome (QTc > 500ms Bazett-formula) and channelopathies that in the opinion of the study PI would significantly compromise participant safety;
* Severe cerebrovascular disorders: cerebral aneurysm or recent/significant stroke;
* Hepatic or renal insufficiency that in the opinion of the Principal Investigator would impact on the ability of the participant to safely participate;
* Narrow angle glaucoma;
* (History of) pheochromocytoma;
* Use of noradrenergic agents;
* Use of CYP2D6 inhibitors (SSRIs, quinidine, terbinafine);
* Use of high dose salbutamol (or other beta2 agonists) that in the opinion of the Principal Investigator would impact on the ability of the participant to safely participate;
* Pregnancy and/or breastfeeding;
* Known hypersensitivity to atomoxetine.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
The percentage of time frozen in the dopaminergic OFF-state | Baseline, visit 2 (one week after baseline) and visit 3 (one week after visit 2).

SECONDARY OUTCOMES:
The percentage of time frozen in the dopaminergic ON-state | Baseline, visit 2 (one week after baseline) and visit 3 (one week after visit 2).
The brain network integration-segregation coefficient | Visit 2 (one week after baseline) and visit 3 (one week after visit 2).